CLINICAL TRIAL: NCT00297778
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Efficacy Study of Pramipexole and Placebo Administered Orally Over a 12 Week Treatment Phase in Parkinson's Disease Patients With Stable Motor Function and Depressive Symptoms
Brief Title: Pramipexole Versus Placebo in Parkinson's Disease (PD) Patients With Depressive Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.596; Eudract 2005-003788-22
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson Disease; Depression
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- pramipexole (Experimental): A daily dose of pramipexole 0.125 mg t.i.d.; titration-to-response up to 1.0 mg t.i.d.
  Interventions: Drug: Pramipexole
- placebo (Placebo Comparator): Placebo (matching) tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pramipexole — Dopamine agonist
  Arms: pramipexole
Other: Placebo
  Arms: placebo

SUMMARY:
Parkinsons Disease (PD) is caused by a decrease of dopamine in a particular part of the brain. Dopamine is a messenger substance (neurotransmitter) that is used by the cells of the brain (nerve cells) to control and harmonize muscle movements. Consequently, the main manifestations of the disease affect movement and include tremor, muscular rigidity, slowness in performing movements and loss of balance.

However, the disease affects also other, non motor functions and may cause other disorders, such as depression. Depression may be a reaction to the disability caused by the disease, but many studies show that depression is more common in PD than in other chronic debilitating illnesses. Moreover, there is also a biological explanation for the phenomenon: dopamine is also used in brain circuits involved in the experience of pleasure, and loss of pleasure in daily physical or social activity is one of the key manifestations of depression.

The objective of the study is to assess whether pramipexole, at doses approved for the treatment of PD symptoms, is more effective than placebo in resolving depressive symptoms in PD patients.

Also data on the safety of the product in the disease will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. 15-item Geriatric Depression Scale (GDS) > or = 5
2. Unified Parkinson's Disease Rating Scale (UPDRS) Part I Score on Question #3 > or = 2
3. Folsteins Mini-Mental State Examination (MMSE) score > 24
4. Male or female patient with PD (UK PD Brain Bank criteria).
5. Patients diagnosed with idiopathic PD, Stage I-III by the Modified Hoehn and Yahr Scale and optimally controlled PD symptoms .
6. Male or female patients aged 30 - 80 years.
7. Ability to provide written informed consent.
8. Women of childbearing potential must have a negative serum beta-humanchoriongonadotropin (Beta-HCG) pregnancy test at the Screening visit unless surgically sterile or last menstruation >or = 12 months prior to signing informed consent.
9. Women of childbearing potential must be using an accepted contraceptive.
10. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Previous history of allergic response, lack of efficacy or complications with pramipexole or its excipients.
2. History of suicidal attempts in the last twelve months; presence of suicidal tendencies/potential.
3. Atypical PD syndromes due to drugs, metabolic disorders, encephalitis or degenerative diseases.
4. History of PD stereotactic brain surgery.
5. Surgery within 180 days of randomization that would negatively impact the patients participation in the study.
6. History of active epilepsy within the past year.
7. Current psychotherapy or behavior therapy while participating the trial
8. Symptomatic orthostatic hypotension prior to randomization.
9. Malignant melanoma or history of previously treated malignant melanoma.
10. Patients who have received typical neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, selegiline or amphetamine derivatives within the past 3 months.
11. Patients who have received dopamine agonists within the past 30 days
12. Electroconvulsive therapy during the 90 days preceding the screening visit (Visit 1).
13. Patients who are currently lactating.
14. Participation in other investigational drug studies or use of other investigational drugs within the previous 30 days prior to randomization.
15. Any other laboratory assay abnormality, which could interfere with patient participation or interpretation of results, or could increase the risk for the patient
16. Any other clinically significant medical/psychiatric condition, which could interfere with patient participation or interpretation of results, or could increase the risk for the patient

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (77):
- Austria (5):
  - 248.596.43003 Boehringer Ingelheim Investigational Site, Graz
  - 248.596.43001 Boehringer Ingelheim Investigational Site, Innsbruck
  - 248.596.43005 Boehringer Ingelheim Investigational Site, Linz
  - 248.596.43004 Boehringer Ingelheim Investigational Site, Sankt Pölten
  - 248.596.43002 Boehringer Ingelheim Investigational Site, Vienna
- 248.596.35801 Boehringer Ingelheim Investigational Site, Oulu, Finland
- France (12):
  - 248.596.3302A Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - 248.596.3302B Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - 248.596.3306A Hôpital Pierre Wertheimer, Bron
  - 248.596.3308A Hôpital Gabriel Montpied, Clermont-Ferrand
  - 248.596.3309A Cabinet Médical, Évreux
  - 248.596.3307A Hôpital Roger Salengro, Lille
  - 248.596.3307B Hôpital Roger Salengro, Lille
  - 248.596.3307C Hôpital Roger Salengro, Lille
  - 248.596.3303A Hôpital La Timone, Marseille
  - 248.596.3305A Hôpital du Haut Levêque, Pessac Cédex
  - 248.596.3305B Hôpital du Haut Levêque, Pessac Cédex
  - 248.596.3301A Hôpital Guillaume et René Laennec, Saint-Herblain
- Germany (11):
  - 248.596.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 248.596.49013 Boehringer Ingelheim Investigational Site, Berlin
  - 248.596.49015 Boehringer Ingelheim Investigational Site, Berlin
  - 248.596.49003 Boehringer Ingelheim Investigational Site, Bremerhaven
  - 248.596.49016 Boehringer Ingelheim Investigational Site, Cologne
  - 248.596.49004 Boehringer Ingelheim Investigational Site, Gera
  - 248.596.49001 Boehringer Ingelheim Investigational Site, Karlsruhe
  - 248.596.49005 Boehringer Ingelheim Investigational Site, Marburg
  - 248.596.49014 Boehringer Ingelheim Investigational Site, Mittweida
  - 248.596.49008 Boehringer Ingelheim Investigational Site, München
  - 248.596.49012 Boehringer Ingelheim Investigational Site, Steglitz
- Italy (8):
  - 248.596.39008 Clinica Neurologica I Policlinico di Catania, Catania
  - 248.596.39004 Neurologia Ospedale della Misericordia, Grosseto
  - 248.596.39005 Clinica Neurologica Policlinico G. Martino, Messina
  - 248.596.39009 Istituti Clinici di Perfezionamento, Milan
  - 248.596.39003 Università degli studi di Napoli "Federico II", Napoli
  - 248.596.39001 Ospedale Civile S. Spirito, Università "G. D'Annunzio", Pescara
  - 248.596.39007 Clinica Neurologica Policlinico Tor Vergata, Roma
  - 248.596.39006 Neurologia Ospedale Evangelico Valdese, Torino
- Netherlands (6):
  - 248.596.31003 Jeroen Bosch Ziekenhuis, locatie WA, 's-Hertogenbosch
  - 248.596.31007 Afdeling neurologie, Amsterdam
  - 248.596.31005 Ziekenhuis Gooi-Noord, Blaricum
  - 248.596.31004 Amphia ziekenhuis, Locatie Molengracht, Breda
  - 248.596.31002 Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - 248.596.31001 Maasland Ziekenhuis, Sittard
- Norway (3):
  - 248.596.47002 Boehringer Ingelheim Investigational Site, Arendal
  - 248.596.47004 Boehringer Ingelheim Investigational Site, Lillehammer
  - 248.596.47003 Boehringer Ingelheim Investigational Site, Sandvika
- Romania (6):
  - 248.596.40003 Boehringer Ingelheim Investigational Site, Bucharest
  - 248.596.40004 Boehringer Ingelheim Investigational Site, Bucharest
  - 248.596.40005 Boehringer Ingelheim Investigational Site, Bucharest
  - 248.596.40001 Boehringer Ingelheim Investigational Site, Cluj-Napoca
  - 248.596.40002 Boehringer Ingelheim Investigational Site, Iași
  - 248.596.40006 Country Clinical Emergency Hospital, Târgu Mureş
- Russia (5):
  - 248.596.70001 Boehringer Ingelheim Investigational Site, Moscow
  - 248.596.70003 Boehringer Ingelheim Investigational Site, Moscow
  - 248.596.70002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 248.596.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 248.596.70005 Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Africa (6):
  - 248.596.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 248.596.27003 Boehringer Ingelheim Investigational Site, Cape Town
  - 248.596.27007 Boehringer Ingelheim Investigational Site, Cape Town
  - 248.596.27008 Boehringer Ingelheim Investigational Site, Johannesburg
  - 248.596.27004 Boehringer Ingelheim Investigational Site, Pretoria
  - 248.596.27006 Boehringer Ingelheim Investigational Site, Richards Bay
- Spain (6):
  - 248.596.34003 Hospital de Alcorcón. Departamento de Neurología, Alcorcon (Madrid)
  - 248.596.34001 Hospital Sta Creu i Sant Pau. Departamento de Neurología, Barcelona
  - 248.596.34002 Hospital Clinic i Provincial. Departamento de Neurología, Barcelona
  - 248.596.34005 Hosp. Univ. Vall d'Hebron. Departamento de Neurología, Barcelona
  - 248.596.34007 Hosp Gral Univ Gregorio Marañón. Departamento de Neurología, Madrid
  - 248.596.34004 Hospital General de Catalunya. Departamento de Neurología, San Cugat Del Valles (Barcelona)
- Sweden (3):
  - 248.596.46004 Boehringer Ingelheim Investigational Site, Linköping
  - 248.596.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 248.596.46002 Boehringer Ingelheim Investigational Site, Stockholm
- Ukraine (5):
  - 248.596.38004 Boehringer Ingelheim Investigational Site, Donetsk
  - 248.596.38005 Boehringer Ingelheim Investigational Site, Kharkiv
  - 248.596.38002 Boehringer Ingelheim Investigational Site, Kiev
  - 248.596.38006 Boehringer Ingelheim Investigational Site, Simferopol
  - 248.596.38003 Boehringer Ingelheim Investigational Site, Vinnytzya

REFERENCES:
- [Derived] Barone P, Poewe W, Albrecht S, Debieuvre C, Massey D, Rascol O, Tolosa E, Weintraub D. Pramipexole for the treatment of depressive symptoms in patients with Parkinson's disease: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2010 Jun;9(6):573-80. doi: 10.1016/S1474-4422(10)70106-X. Epub 2010 May 7. PMID 20452823
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/248/248.596_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet matching active treatment
- Pramipexole: Ascending dose titration of Pramipexole. Pramipexole doses consisted of 0.125 mg three times daily (t.i.d), 0.25mg t.i.d, 0.5mg, t.i.d, 0.25mg+0.5mg t.i.d and 1.0 mg t.i.d.
Period: Overall Study
Arm/Group | Placebo | Pramipexole
Started | 152 | 144
Completed | 133 | 124
Not Completed | 19 | 20
Not completed — Adverse Event | 16 | 10
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lack of Efficacy | 2 | 1
Not completed — Non-compliant with trial protocol | 0 | 3
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pramipexole | Total
Number analyzed (Participants) | 152 | 144 | 296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (9.9) | 67.4 (9.0) | 67 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 82 | 156
  Male | 78 | 62 | 140

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Beck Depression Inventory-Version 1A (BDI-IA) Total Score at Week 12
Description: The BDI measures symptoms of depression on an ordinal scale ranging from 0 (no symptoms) to 63 (worst symptoms)
Time Frame: Baseline and Week 12
Population: The Full analysis set (FAS) made up of all randomised and treated participants with a baseline and at least one on-treatment assessment of the BDI. 9 participants from those randomised and treated were excluded due to insufficient BDI data.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
Score on scale | -4 (0.5) | -5.9 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.0103, ANCOVA; Mean Difference (Net) = -1.9, 95% CI [-3.4 to -0.5]

2. Secondary Outcome: Change in BDI-IA Clinical Response (at Least 50% Reduction in Symptoms) at Week 12
Description: BDI clinical response was defined as a reduction of ≥50% from baseline
Time Frame: Week 12
Population: FAS. 10 participants from those randomised and treated were excluded due to insufficient BDI data (1 due to a zero baseline score).
Measure: Number; unit: participants
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 147 | 139
participants | 27 | 38
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.0535, Regression, Logistic; Odds Ratio (OR) = 1.758, 95% CI [0.992 to 3.115]

3. Secondary Outcome: Change From Baseline in the Geriatric Depression Scale-Short Form (GDS-SF) (15-item Version) Total Score at Week 12
Description: The GDS measures symptoms of depression on an ordinal scale ranging from 0 (no symptoms) to 15 (worst symptoms)
Time Frame: Baseline and Week 12
Population: FAS. 9 participants from those randomised and treated were excluded due to insufficient GDS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
units on a scale | -1.7 (0.3) | -2.5 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.0346, ANCOVA; Mean Difference (Net) = -0.8, 95% CI [-1.5 to -0.1]

4. Secondary Outcome: Change From Baseline in Snaith-Hamilton Pleasure Scale (SHAPS) Total Score at Week 12
Description: The SHAPS measures anhedonia (inability to experience pleasure) on an ordinal scale ranging from 0 (no anhedonia) to 14 (worst anhedonia)
Time Frame: Baseline and Week 12
Population: FAS. 9 participants from those randomised and treated were excluded due to insufficient SHAPS data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
units on a scale | 0 [-2 to 0] | 0 [-2 to 0]
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.5244, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0, 95% CI [-1 to 0]

5. Secondary Outcome: Change From Baseline in the Unified Parkinson's Disease Rating Scale (UPDRS) Part I Depression Score at Week 12
Description: The UPDRS part I depression score measures depression on an ordinal scale ranging from 0 (none) to 4 (sustained depression/suicidal thoughts)
Time Frame: Baseline and Week 12
Population: FAS. 9 participants from those randomised and treated were excluded due to insufficient UPDRS data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
units on a scale | -1 [-1 to 0] | -1 [-2 to 0]
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.141, van Elteren (country stratification); Median Difference (Net) = 0, 95% CI [0 to 0]

6. Secondary Outcome: Change From Baseline in the UPDRS Part II Total Score at Week 12
Description: Unified Parkinson's Disease Rating Scale part II total score on FAS The UPDRS part II total score measures the impact of PD on activities of daily living on an ordinal scale ranging from 0 (normal) to 52 (worst symptoms)
Time Frame: Baseline and Week 12
Population: FAS. 9 participants from those randomised and treated were excluded due to insufficient UPDRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
units on a scale | -1.2 (0.3) | -2.4 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Net) = -1.2, 95% CI [-1.9 to -0.4]

7. Secondary Outcome: Change From Baseline in the UPDRS Part III Total Score at Week 12
Description: The UPDRS part III total score measures the impact of PD on motor skills on an ordinal scale ranging from 0 (normal) to 108 (worst symptoms)
Time Frame: Baseline and Week 12
Population: FAS. 10 participants from those randomised and treated were excluded due to insufficient UPDRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 138
units on a scale | -2.2 (0.5) | -4.4 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.0034, ANCOVA; Mean Difference (Net) = -2.2, 95% CI [-3.7 to -0.7]

8. Secondary Outcome: Change From Baseline in the UPDRS Part II+III Total Score at Week 12
Description: The UPDRS part II+III total score measures the impact of PD on activities of daily living and motor skills on an ordinal scale ranging from 0 (normal) to 160 (worst symptoms)
Time Frame: Baseline and Week 12
Population: FAS. 10 participants from those randomised and treated were excluded due to insufficient UPDRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 138
units on a scale | -3.4 (0.7) | -6.8 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Net) = -3.4, 95% CI [-5.4 to -1.5]

9. Secondary Outcome: Clinical Global Impressions of Global Improvement (CGI-I) at Week 12
Description: The CGI-I measures the overall improvement in the participants condition from baseline on an ordinal scale ranging from 1 (very much improved) to 7 (very much worse)
Time Frame: Week 12
Population: FAS. 9 participants from those randomised and treated were excluded due to insufficient CGI-I data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
units on a scale | 3 [1 to 6] | 3 [1 to 6]
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.821, 95% CI [1.187 to 2.794]

10. Secondary Outcome: Change From Baseline in the Parkinson's Disease Questionnaire-39 (PDQ-39) Overall Index Score at Week 12
Description: The PDQ-39 measures aspects of health in PD participants, the overall index score is the mean of the eight individual domain scores measured on a continuous scale ranging from 0 (no problem at all) to 100 (maximum level of the problem)
Time Frame: Baseline and Week 12
Population: FAS. 52 participants from those randomised and treated were excluded due to insufficient PDQ-39 data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 127 | 108
units on a scale | -2.4 [-8.9 to 2.6] | -3.3 [-8.9 to 0.3]
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.1925, van Elteren (country stratification); Median Difference (Net) = -1.3, 95% CI [-3.3 to 0.8]

11. Secondary Outcome: Change From Baseline in the European Quality of Life Scale (EUROQOL (EQ)-5D) Overall Index Score at Week 12
Description: This is a 5-item patient reported measure of health status developed for use in evaluating health and healthcare. It produces a numeric score for health status on which full health has a value of 1 and death has a value of 0. Euro-QOL describes health status in terms of 5 dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. The EQ-5D measures health status on a continuous scale ranging from 0 (dead) to 1 (full health)
Time Frame: Baseline and Week 12
Population: FAS. 16 participants from those randomised and treated were excluded due to insufficient EQ-5D data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 144 | 136
units on a scale | 0 [-0.06 to 0.12] | 0.07 [0 to 0.21]
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.0337, Wilcoxon rank sum (Van Elteren's test); Hodges-Lehmann est of diff in medians = 0.04, 95% CI [0 to 0.09]

12. Secondary Outcome: Change From Baseline to End of Maintenance Phase in European Quality of Life Visual Analogue Scale (EUROQOL (EQ) VAS) Pain Score at Week 12
Description: The VAS is a method used for the measurement of pain. The patient is asked to place a mark on an uncalibrated (usually 0 - 10 cm) line representing the patient's degree of general pain. The two extremities of the line were taken to represent 'no pain' and 'unbearable pain', respectively. VAS pain scores could range from 0 (no pain) to 100 (unbearable pain).
Time Frame: Baseline and Week 12
Population: FAS. 15 participants from those randomised and treated were excluded due to insufficient EQ-5D data.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
mm | -3 (1.8) | -3.5 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; Test type: Superiority or Other; p = 0.8471, ANCOVA; Mean Difference (Net) = -0.5, 95% CI [-5.6 to 4.6]

13. Secondary Outcome: Change From Baseline in the UPDRS Part I Total Score at Week 12
Description: The UPDRS part I total score measures depression on an ordinal scale ranging from 0 to 16. UPDRS Part I total scores could range from 0 to 16; where higher scores were indicative of worse symptoms.
Time Frame: Baseline and Week 12
Population: FAS. 9 participants from those randomised and treated were excluded due to insufficient UPDRS data.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 148 | 139
units on a scale | -1.0 [-1.0 to 0.0] | -1.0 [-2.0 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; N's exclude patients from the analysis set with incomplete data; Test type: Superiority or Other; p = 0.1410, Wilcoxon rank sum (Van Elteren's test); Hodges-Lehmann est of diff in medians = 0.0, 95% CI 2-sided [0.0 to 0.0] — 95% Confidence interval is Distribution-free Confidence Interval (Moses)

14. Secondary Outcome: Change From Baseline in the UPDRS Part IV Total Score at Week 12
Description: The UPDRS Part IV measures motor complications (dyskinesia) and the total score could range from 0 to 23; where higher scores were indicative of worse symptoms.
Time Frame: Baseline and Week 12
Population: FAS. 28 participants from those randomised and treated were excluded due to insufficient UPDRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 137 | 131
units on a scale | -0.2 (0.1) | -0.3 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Pramipexole; N's exclude patients from the analysis set with incomplete data; Test type: Superiority or Other; p = 0.5231, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.2

15. Secondary Outcome: Abnormal Findings: Clinical Laboratory Evaluations (Biochemistry and Haematology)and Vital Signs
Time Frame: Baseline and Week 12
Measure: Number; unit: participants
Arm/Group | Placebo | Pramipexole
Number analyzed (Participants) | 152 | 144
participants
  Hypotension | 1 | 1
  Orthostatic hypotension | 1 | 0

ADVERSE EVENTS:
Time Frame: First drug intake up to 48 hours after the last drug intake
Arm/Group | Placebo | Pramipexole
Serious Adverse Events (participants affected / at risk) | 6 | 6
Other Adverse Events (participants affected / at risk) | 58 | 71
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | Pramipexole
Endocarditis (Infections and infestations) | 0/152 | 1/144
Hyperlipidaemia (Metabolism and nutrition disorders) | 0/152 | 1/144
Hallucination (Psychiatric disorders) | 0/152 | 1/144
Cerebral haemorrhage (Nervous system disorders) | 0/152 | 1/144
Cerebrovascular accident (Nervous system disorders) | 0/152 | 1/144
Parkinson disease (Nervous system disorders) | 1/152 | 0/144
Radicular pain (Nervous system disorders) | 1/152 | 0/144
Syncope (Nervous system disorders) | 0/152 | 1/144
Angina unstable (Cardiac disorders) | 1/152 | 0/144
Cardiac failure (Cardiac disorders) | 1/152 | 1/144
Abdominal pain (Gastrointestinal disorders) | 1/152 | 0/144
Gastroduodenal ulcer (Gastrointestinal disorders) | 1/152 | 0/144
Volvulus (Gastrointestinal disorders) | 1/152 | 0/144
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/152 | 1/144
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/152 | 0/144
Anuria (Renal and urinary disorders) | 0/152 | 1/144
Accident at home (Injury, poisoning and procedural complications) | 1/152 | 0/144
Comminuted fracture (Injury, poisoning and procedural complications) | 1/152 | 0/144
Fall (Injury, poisoning and procedural complications) | 1/152 | 1/144
Femoral neck fracture (Injury, poisoning and procedural complications) | 0/152 | 1/144
Skull fracture base (Injury, poisoning and procedural complications) | 1/152 | 0/144
Traumatic brain injury (Injury, poisoning and procedural complications) | 1/152 | 0/144
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo | Pramipexole
Insomnia (Psychiatric disorders) | 4/152 | 8/144
Dizziness (Nervous system disorders) | 9/152 | 16/144
Headache (Nervous system disorders) | 12/152 | 16/144
Somnolence (Nervous system disorders) | 12/152 | 15/144
Dyskinesia (Nervous system disorders) | 4/152 | 10/144
Vertigo (Ear and labyrinth disorders) | 4/152 | 10/144
Nausea (Gastrointestinal disorders) | 26/152 | 24/144
Fatigue (General disorders) | 9/152 | 8/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.